CLINICAL TRIAL: NCT04274647
Title: Skin Sensitization Test (Modified Draize-95) to Support a Low Dermatitis Potential Claim
Brief Title: Skin Sensitization Test (Modified Draize-95 Test)
Acronym: Draize-95
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YTY Industry (Manjung) Sdn Bhd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-MDT-02-17-19
Record Dates: First submitted 2020-02-17; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2019-07

CONDITIONS: Skin Sensitisation

STUDY DESIGN:
Intervention Model Description: NON-STERILE, POWDER FREE NITRILE EXAMINATION GLOVES, LOW DERMATITIS POTENTIAL, TESTED FOR USE WITH CHEMOTHERAPY DRUGS - BLUE
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device and Control (Experimental): NON-STERILE, POWDER FREE NITRILE EXAMINATION GLOVES, LOW DERMATITIS POTENTIAL, TESTED FOR USE WITH CHEMOTHERAPY DRUGS - BLUE Approximately 2cm x 2cm square positioned to ensure that the inside portion of the test material maintained skin contact.
  Positive control: 0.4% sodium lauryl sulfate (SLS) Dose. 0.2ml
  Interventions: Device: NON-STERILE, POWDER FREE NITRILE EXAMINATION GLOVES, LOW DERMATITIS POTENTIAL, TESTED FOR USE WITH CHEMOTHERAPY DRUGS - BLUE

INTERVENTIONS:
Device: NON-STERILE, POWDER FREE NITRILE EXAMINATION GLOVES, LOW DERMATITIS POTENTIAL, TESTED FOR USE WITH CHEMOTHERAPY DRUGS - BLUE — Approximately 2cm x 2cm square positioned to ensure that the inside portion of the test material maintained skin contact.

SUMMARY:
Skin Sensitization Test (Modified Draize-95) to Support a Low Dermatitis Potential Claim for a Blue Non Sterile Powder Free Nitrile Examination Gloves. To evaluate whether residual chemical additives at a level that may induce type IV allergy in the unsensitized general user population are present in a finished rubber containing medical device.

DETAILED DESCRIPTION:
1. To evaluate whether residual chemical additives at a level that may induce Type IV allergy in the unsensitized general user population are present in a finished rubber containing medical device.
2. To meet requirements for claim: This product demonstrated reduced potential for sensitizing users to chemical additives as described in Guidance for Industry and FDA Staff - Medical Glove Guidance Manual9. Supporting Test Data: A negative skin sensitization test (Modified Draize-95 Test) on a minimum of 200 non-sensitized human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be aged 18 and 65 years, inclusive;
* Subjects who have not participated in other voluntary testing for at least 30 days;
* Subjects must be capable of understanding and following directions.
* Female subjects must produce a negative urine pregnancy test prior to the initiation and also at the completion of the tiral.

Exclusion Criteria:

* Subjects who are in ill health;
* Subjects who are taking medication, other than birth control, which could influence the purpose, integrity or outcome of the tiral;
* Subjects who have used topical or systemic corticosteriods, anti-inflammatories, antihistamines or antibiotics within 2 weeks prior to trial initiationor during their participation on this tiral;
* Femable subjects who are pregnant as evidenced by a urine pregnancy test, planning to become pregnant or lactaticn during the tiral;
* Subjects who have a history of adverse reactions to cosmetics, OTC drugs, or other personal care products;
* Subjects who introduce the use of any new cosmetic, toiletry or personal care products during the trial;
* Subjects with any visible skin disease that might be confuesd with skin reactions caused by the test material;
* Subjects with any knowledge or indication of existing Type IV allergy (delayed hypersensitivity) to natural rubber chemical additives;
* Subjects with a history of frequent irritation; or
* Subjects who have received endogenious or exogenious immunosuppressive treatment (r prolonged exposure to sun).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 208 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Irritation scored by Erythemal Scoring Scale | 8 weeks
  0 - No visible reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Samy, Sitiawan, Perak, Malaysia